CLINICAL TRIAL: NCT00110201
Title: Prophylactic Use of Nesiritide (Brain Natriuretic Peptide, BNP) for the Prevention of Acute Renal Failure in Thoracic Aortic Aneurysm Surgery Patients
Brief Title: The Use of Nesiritide in Thoracic Aneurysm Repair to Prevent Acute Renal Failure
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ejaz, Abulate A, MD (Individual)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: bnpufl2005; 20050059
Record Dates: First submitted 2005-05-04; First posted 2005-05-05 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2005-05

CONDITIONS: Cardiovascular Disease; Acute Renal Failure; Death
Keywords: Acute renal failure; Nesiritide; Cardiovascular surgery
MeSH Terms: conditions — Cardiovascular Diseases; Acute Kidney Injury; Death | interventions — Natriuretic Peptide, Brain

INTERVENTIONS:
Drug: Nesiritide

SUMMARY:
The purpose of this trial is to study the use of nesiritide in thoracic aneurysm repair to prevent acute renal failure.

The study hypothesis: Nesiritide, given prophylactically prior to surgery may prevent acute renal failure requiring dialysis and/or decrease mortality.

DETAILED DESCRIPTION:
Acute renal failure is a major and serious complication of more than 200,000 cardiovascular surgeries performed on adult Americans annually (www.sts.org). The incidence of acute renal failure (ARF) after cardiac surgery (depending on criteria used to define ARF) is 1-5%, in the absence of preexisting renal dysfunction. The subset of patients with thoracic aortic aneurysm surgery have a higher risk for the development of postoperative ARF (25-40% - ARF defined as doubling of serum creatinine; 13% - ARF defined as requirement for dialysis). This risk is further increased by various peri-operative factors, especially cardiopulmonary bypass time.

The overall postoperative mortality rate for cardiovascular surgery is 2.2%, but is much higher for thoracic aortic aneurysm surgery (8-10% for elective repair, 25-50% for ruptured thoracic aorta aneurysm repair). The major risk factor for thoracic aortic aneurysm surgery related mortality is post-operative ARF requiring dialysis. When thoracic aortic aneurysm surgery is complicated by acute renal failure, the mortality rate worsens to 50%. Thus, identifying ways to prevent acute renal failure may have a major impact on the outcome of cardiovascular surgery. A retrospective study of the use of nesiritide in cardiovascular surgery patients by our group has demonstrated a tendency towards a decreased incidence of renal failure and mortality, when the medication is used prophylactically.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Undergoing thoracic aortic aneurysm surgery
* Impaired renal function

Exclusion Criteria:

* Prior history of allergy/adverse reaction to Nesiritide
* History of any organ transplant
* Preoperative intra-aortic balloon pump (IABP)
* Decompensated congestive heart failure (CHF)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124
Dates: Start 2005-03; Study Completion 2007-12

PRIMARY OUTCOMES:
Need for dialysis and/or mortality

SECONDARY OUTCOMES:
Rise in serum creatinine
blood urea nitrogen

CONTACTS AND LOCATIONS:
Locations (1):
- Shands Hospital at the University of Florida, Gainesville, Florida, United States

REFERENCES:
- [Derived] Hashimoto H, Yamada H, Murata M, Watanabe N. Diuretics for preventing and treating acute kidney injury. Cochrane Database Syst Rev. 2025 Jan 29;1(1):CD014937. doi: 10.1002/14651858.CD014937.pub2. PMID 39878152
- [Derived] Dass B, Shimada M, Kambhampati G, Ejaz NI, Arif AA, Ejaz AA. Fluid balance as an early indicator of acute kidney injury in CV surgery. Clin Nephrol. 2012 Jun;77(6):438-44. doi: 10.5414/cn107278. PMID 22595385
- [Derived] Ejaz AA, Beaver TM, Shimada M, Sood P, Lingegowda V, Schold JD, Kim T, Johnson RJ. Uric acid: a novel risk factor for acute kidney injury in high-risk cardiac surgery patients? Am J Nephrol. 2009;30(5):425-9. doi: 10.1159/000238824. Epub 2009 Sep 11. PMID 19752530
- [Derived] Ejaz AA, Martin TD, Johnson RJ, Winterstein AG, Klodell CT, Hess PJ Jr, Ali AK, Whidden EM, Staples NL, Alexander JA, House-Fancher MA, Beaver TM. Prophylactic nesiritide does not prevent dialysis or all-cause mortality in patients undergoing high-risk cardiac surgery. J Thorac Cardiovasc Surg. 2009 Oct;138(4):959-64. doi: 10.1016/j.jtcvs.2009.05.014. Epub 2009 Jul 3. PMID 19660420